CLINICAL TRIAL: NCT00798421
Title: Pilot Study to Develop a Model to Evaluate Nosocomial Transmission of Influenza
Brief Title: Study to Evaluate Nosocomial Transmission of Influenza
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Iain Stephenson, University of Leicester, UK
Other Study IDs: UHL10421; REC 07/H0402/59
Record Dates: First submitted 2008-11-25; First posted 2008-11-26 (Estimated); Last update posted 2008-11-26 (Estimated); Status verified 2008-11

CONDITIONS: Influenza
Keywords: Influenza, transmission
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Throat and nose swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Heathcare worker: health care worker exposed to patient with influenza

SUMMARY:
The purpose of this study is to investigate whether influenza can be reliably transmitted from children to susceptible contacts in a health care setting. The goal is to develop a transmission that can then be used to assess interventions to prevent transmission

Research objectives:

To develop a model to investigate the frequency of influenza transmission from an infected child to a susceptible health care worker

Research Hypotheses:

Influenza viruses can be transmitted from infected children to exposed health care workers

DETAILED DESCRIPTION:
CHildren with influenza infection presenting to ED will be identified by RAT. Healthy healthcare worker subjects will expose themselves and perform specific activities with the child.

subjects will be followed by diary card, clinical symptom scores and virology swabs to assess frequency of transmission

ELIGIBILITY:
Inclusion criteria:

* Infected Children

  * Age < 16 years
  * Parents or legal guardians willing to give informed written consent
  * Presenting with a febrile illness confirmed as influenza by near patient rapid antigen testing
* Healthy volunteers

  * Willing to give informed written consent

Exclusion criteria

* Children

  * No parents or legal guardians able to give informed consent
* Healthy volunteers

  * known allergy to oseltamivir or zanamivir
  * presence of underlying condition or concomitant therapy requiring dose alteration of oseltamivir (severe renal or hepatic failure; methotrexate and probenecid)
  * underlying immunosuppressive disorder
  * known galactose intolerance
  * underlying chronic medical condition known to increase risk of influenza-related complications (including asthma, chronic pulmonary airways disease, chronic cardiovascular disease, diabetes mellitus, chronic neurological disorder)
  * inability or contraindication to collection of nasal swabs
  * previous influenza vaccination within 2 years
  * current smoker
  * pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Healthy subject volunteers > 18 years of age
  2. Children with confirmed influenza presenting to the Children's Hospital, Leicester Royal Infirmary
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-04 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of transmission of influenza | 1 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Iain Stephenson, FRCP, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals Leicester, Leicester, Leics, United Kingdom